CLINICAL TRIAL: NCT00222911
Title: Conservative Treatment of Plantar Fasciitis With Dorsiflexion Night Splints and Medial Arch Supports: a Prospective Randomized Study
Brief Title: Treatment of Plantar Fasciitis With Dorsiflexion Night Splints and Medial Arch Supports
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Saudi Arabian Cultural Mission (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0506173
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2008-05-20 (Estimated); Status verified 2008-05

CONDITIONS: Plantar Fasciitis
Keywords: plantar fasciitis; heel pain; heel spur; night splint; arch support; foot orthosis; physical therapy
MeSH Terms: conditions — Fasciitis, Plantar; Heel Spur

INTERVENTIONS:
Device: dorsiflexion night splint
Device: medial arch support

SUMMARY:
The overall purpose of this study is to examine the combined effect of both dorsiflexion night splints and medial arch supports and compare it to the effect of these interventions each by itself in the treatment of plantar fasciitis.

DETAILED DESCRIPTION:
Plantar fasciitis is an overuse injury causing inflammation at the origin of the plantar fascia and is characterized by plantar heel pain that is provoked by taking the first few steps in the morning and by prolonged standing. It is the most common clinical problem that causes inferomedial heel pain in adults. It is estimated that more than two million people receive treatment for plantar fasciitis in the United States each year. Despite its familiarity to physicians, the exact etiology of plantar fasciitis remains obscure. The variety of treatments noted in the literature attests to the uncertainty of the etiology and pathogenesis of plantar fasciitis. It has been suggested that the success of conservative care for the treatment of patients with plantar fasciitis requires a combination of treatment modalities. Although many authors have stated that mechanical therapy should be considered a cornerstone of any effective treatment plan, some debate remains regarding the most effective form of mechanical treatment. The literature provides evidence to support the use of dorsiflexion night splints and medial arch supports in the treatment of plantar fasciitis. A night splint is used to address early morning pain by preventing contracture of the plantar fascia and Achilles tendon overnight. An arch support, on the other hand, addresses the end of the day pain by preventing overstretch of the plantar fascia during prolonged weight bearing. Therefore, both night splints and arch supports may be necessary to treat plantar fasciitis as they complement each other by both controlling nocturnal contracture of the plantar fascia and Achilles tendon and reducing stresses imposed on the plantar fascia during the day, respectively. This prospective randomized study, to the best of our awareness, is the first that addresses this problem by examining the combined effect of these treatment modalities and comparing it to the effect of a night splint or arch support each by itself. We hypothesize that the night splint and arch support together will be more effective in the treatment of plantar fasciitis than night splint or arch support alone in terms of increasing the range of pain-free passive ankle dorsiflexion, relieving heel tenderness and pain, and reducing disability imposed by the heel pain/plantar fasciitis. A secondary hypothesis of this study is that those with limited passive dorsiflexion of the ankle will benefit from a night splint more than those with normal passive dorsiflexion of the ankle and those with a low medial longitudinal arch will benefit from an arch support more than those with a normal medial longitudinal arch in terms of the previously mentioned outcomes. The range of motion will be measured with a goniometer; heel tenderness will be measured with a pressure algometer; and pain and disability will be measured by the Foot Function Index.

ELIGIBILITY:
Inclusion Criteria:

* plantar heel pain
* pain is provoked by taking the first few steps in the morning, by standing after prolonged sitting, and/or by prolonged standing
* tenderness localized to the origin of the plantar fascia on the medial calcaneal tubercle

Exclusion Criteria:

* previous foot surgery
* foot trauma within the previous three months
* tarsal tunnel syndrome
* loss of plantar foot sensation
* foot pathology other than plantar fasciitis including tendonitis, bursitis, or calcaneus fracture
* generalized inflammatory disorders associated with the diagnosis of plantar fasciitis including rheumatoid arthritis, ankylosing spondylitis, Reiter's disease, gout, or lupus
* previous treatment of plantar fasciitis with dorsiflexion night splints and/or medial arch supports
* inability or unwillingness to discontinue current treatment modalities that are used for the purpose of plantar fasciitis
* participation in a worker's compensation program
* age of less than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2005-08; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
the range of pain-free passive ankle joint dorsiflexion at baseline and 6 weeks
plantar heel tenderness at baseline and 6 weeks
plantar heel pain at baseline and 6 weeks
disability imposed by the heel pain/plantar fasciitis at baseline and 6 weeks

SECONDARY OUTCOMES:
medial longitudinal arch height at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad H Alghadir, MS, PT, Principal Investigator — University of Pittsburgh; James Irrgang, PhD, PT, Study Chair — University of Pittsburgh; Anthony Delitto, PhD, PT, Study Director — University of Pittsburgh; Dane Wukich, MD, Study Director — University of Pittsburgh; Ray Burdett, PhD, PT, Study Director — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States